CLINICAL TRIAL: NCT06012968
Title: Study on the Protective Effect of Gastrodin on Myocardial Injury in Patients Undergoing Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: mzk202301
Record Dates: First submitted 2023-08-20; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GAS
- Control

SUMMARY:
This study intends to include hypertrophic cardiomyopathy patients over 18 years old who underwent cardiac surgery in our hospital. Patients were divided into medication group and control group according to the use of gastrodin during operation. The patients ' myocardial tissue samples were collected, the postoperative prognosis data were observed and recorded, and the data were analyzed. The degree of myocardial tissue cell damage and postoperative clinical outcomes were compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypertrophic cardiomyopathy aged≥18 years, regardless of gender;
* Patients undergoing elective hypertrophic cardiomyopathy outflow tract surgery;
* Signed informed consent, good compliance.

Exclusion Criteria:

* suffering from more serious genetic diseases (such as immunodeficiency, thalassemia, etc.);
* moderate to severe malnutrition, moderate to severe anemia;
* persistent infection;
* severe preoperative underlying diseases (such as severe liver and kidney dysfunction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients included in this study were preoperatively diagnosed as hypertrophic cardiomyopathy.
  Diagnosis of hypertrophic cardiomyopathy: according to the medical history and physical examination, echocardiography showed diastolic ventricular septal thickness of 15 mm.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Degree of myocardial cell injury | During postoperative hospitalization stay, an average of about two weeks
  Postoperative myocardial injury marker serum concentration, postoperative cardiac function ultrasound index

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China